CLINICAL TRIAL: NCT02875678
Title: A Single-Dose Study to Evaluate the Effects of ABX-1431 on Gastric Accommodation and Nutrient Volume Tolerance in Patients With Functional Dyspepsia
Brief Title: A Study to Evaluate the Effects of ABX-1431 on Patients With Functional Dyspepsia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: Abide Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ABX-1431_PN005
Record Dates: First submitted 2016-07-13; First posted 2016-08-23 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — ABX-1431

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABX-1431 (Experimental): ABX-1431, capsules, 40 mg, single dose
  Interventions: Drug: ABX-1431
- Placebo (Placebo Comparator): Placebo, capsules, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX-1431 — Single-dose ABX-1431
  Arms: ABX-1431
Drug: Placebo — Single-dose matching placebo
  Arms: Placebo

SUMMARY:
A Single-Dose Study to Evaluate the Effects of ABX-1431 on Gastric Accommodation and Nutrient Volume Tolerance in Patients with Functional Dyspepsia.

DETAILED DESCRIPTION:
This is a single dose, randomized, placebo-controlled, two period crossover study. This study will assess the effects of ABX-1431 on gastric physiology in patients with functional dyspepsia, who have clinical evidence of impaired gastric accommodation with meals.

All patients will undergo a screening visit for enrollment criteria. Eligible patients will be treated with a single dose of ABX-1431 HCl or placebo followed by IGP measurement, measured with a high resolution manometry probe during a nutrient volume tolerance test. After a washout period of at least one week, patients will undergo identical procedures with the other treatment.

This study will enroll 12 functional dyspepsia (FD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has functional dyspepsia, postprandial distress syndrome (PDS) subtype, defined by the Rome III criteria.
* Patient has evidence of impaired gastric accommodation.
* Patient's Rome III Questionnaire results indicates that the intensity of co-existing epigastric pain and/or epigastric burning may be present, but have the same or lesser intensity than the evaluations of postprandial fullness or early satiety (i.e. epigastric pain and burning are not the prominent symptoms of the patient's functional dyspepsia).
* Patient recall of symptoms of gastrointestinal reflux over the past 8 weeks has no more than 2 episodes per week of heartburn or regurgitation.
* Patient is a male or female between 18 and 65 years of age at the pre-study/screening visit.
* Patient has a Body Mass Index (BMI) >18 to ≤30 kg/m2 at the pre-study/screening visit.
* Patient is judged to have no unmanaged significant disease or disorder based on medical history, physical examination, vital sign measurements, and laboratory safety obtained at pre-study/screening, and within 36 hours prior to first administration of study drug.
* Patient has no clinically significant abnormality of ECG performed at pre study/screening, and prior to first administration of study drug.
* Patient is willing to undergo the nutrient volume tolerance tests.

Exclusion Criteria:

* Patient is under the age of legal consent.
* Female patients who are pregnant or breastfeeding.
* Patient has a personal history of a clinically significant psychiatric disorder (including severe affective disorder, anxiety disorder, post-traumatic stress disorder, psychotic disorder or drug-induced psychoses).
* Patient has a first-degree family history of schizophrenia, severe affective disorder, severe anxiety disorder, or other psychosis.
* Patient is taking antidepressants including SSRIs, SNRIs, tricyclic antidepressants, or atypical antidepressant medications such as bupropion, mirtazapine, trazodone or agomelatine. Patients taking these or other types of medicine for anxiety are also excluded. Patients who have discontinued antidepressants more than 6 months ago may be enrolled at the discretion of the Investigator. Patients who are taking gabapentin or pregabalin or buspirone are also excluded.
* Patient is mentally or legally incapacitated, has significant emotional problems at the time of pre-study/screening visit or is expected to have potential for mental incapacitation during the conduct of the study.
* Patient has had any gastrointestinal surgery. Those having undergone a simple appendectomy more than 1 year prior to the pre-study/screening visit may participate.
* Patient has had any acute gastrointestinal illness in the past 3 months.
* Patient has laboratory tests at screening or within 36 hours of first administration of study drug outside of these limits: Aspartate transaminase (AST) >1.5 x upper limit of normal (ULN) or Alanine transaminase (ALT) >1.5 x ULN.
* Patient has an estimated creatinine clearance (CrCl) of ≤80 mL/min based on the Cockcroft-Gault equation. An actual creatinine clearance, as measured using a 24-hour urine collection, may be used in place of, or in conjunction with the Cockcraft-Gault calculation. Patients with an actual or calculated creatinine clearance that is in the range of 72-79 mL/min (i.e., within 10% of 80 mL/min) may be enrolled in the study at the discretion of the Investigator.
* Patient has an active or prior history of neurological disorder, including but not limited to seizure disorder, epilepsy, stroke, neurological disease, cognitive impairment, head trauma with prolonged loss of consciousness (>10 minutes), or migraine headaches.
* Patient has a history of clinically significant neoplastic disease, with the exception of adequately treated localized or in situ non-melanoma carcinoma of the skin (e.g., basal cell carcinoma) or the cervix.
* Patient has a family history of long QT syndrome.
* Patient has a QTc interval of >450 msec (male patients) or >470 msec (female patients).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Difference from placebo in area above the curve of intragastric pressure (mm Hg) during a liquid meal infusion on Day 1 | Through Day 1 of dosing

SECONDARY OUTCOMES:
Difference from placebo in nutrient volume tolerance (ml) on Day 1 placebo. | Through Day 1 of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Chan Beals, MD,PhD, Study Director — Abide Therapeutics
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided